CLINICAL TRIAL: NCT02847806
Title: Effects of Replacement Therapy With Sexual Steroid Hormones on the Insulin Sensitivity of Hypogonadal Man
Acronym: STEROSENS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 07-034
Record Dates: First submitted 2015-08-13; First posted 2016-07-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-07

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Estradiol; Insulin; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol (Experimental): dosage used in the study: 1 patch / 3-4 days dosed at 25, 37.5 or 50 mg / 24h titration according to the plasma level, with the objective of a physiological level of estradiol (25-40 pg / ml ) - During 4 weeks
  Interventions: Biological: Estradiol (Insulin sensitivity)
- Testosterone (Experimental): dosage used : from 25 to 75 mg / day of testosterone (ie 2.5 to 7.5 g / day transdermal gel) according to the plasma level, with the goal of a physiological level of testosterone (5-8 ng / ml) - During 4 weeks
  Interventions: Biological: Testosterone (Insulin sensitivity)
- Testosterone + Estradiol (Experimental): Testosterone + Estradiol During 4 weeks
  Interventions: Biological: Estradiol (Insulin sensitivity); Biological: Testosterone (Insulin sensitivity)

INTERVENTIONS:
Biological: Estradiol (Insulin sensitivity)
  Arms: Estradiol; Testosterone + Estradiol
Biological: Testosterone (Insulin sensitivity)
  Arms: Testosterone; Testosterone + Estradiol

SUMMARY:
Sexual steroids administered to supra-physiological doses are likely to change the carbohydrate and lipid metabolism.

Investigators propose to study in 12 hypogonadal men hypogonadotropic or hypergonadotropic treated with aromatase inhibitor, the respective effects of estradiol, testosterone or both steroids administered in a cross-over Latin squares plan on insulin sensitivity measured by the reference method of the hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadism hypogonadotropic or hypergonadotropic
* Man aged 18-60 years
* BMI between 18 and 27.

Exclusion Criteria:

* Other ante-pituitary deficiency
* Chronic treatment modifying carbohydrate metabolism (thiazides, beta 2 mimetics, steroids ...)
* Diabetes
* Obesity diffuse or android
* Hemochromatosis
* osteoporosis
* chronic diseases
* neoplasia
* High blood pressure

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
GIR (glucose infusion rate) during euglycemic hyperinsulinemic clamp | change between baseline and after 4 weeks of treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Unit and Clinical Research Center Basse Normandie, University Hospital of Caen, Caen, France